CLINICAL TRIAL: NCT04009915
Title: Comparison of Curative Effect and Postoperative Survival Rate Between Video-assisted Thoracoscopic Surgery and Open Thoracic Surgery for Stage II - III Lung Cancer, A Prospective, Randomized, Controlled Trial: (The VOLCANO Study)
Brief Title: VATS VS. Open Thoracic Surgery for Stage II - III Lung Cancer
Acronym: VOLCANO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, duan liang, Principal Investigator, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Duanliang 1
Record Dates: First submitted 2019-07-03; First posted 2019-07-05 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer; Surgery
MeSH Terms: conditions — Lung Neoplasms | interventions — Thoracic Surgery, Video-Assisted; Conversion to Open Surgery

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VATS (Experimental): Patients undergo a standard VATS operation for stage II-III lung cancer
  Interventions: Procedure: VATS
- open surgery (Active Comparator): Patients undergo a standard open operation for stage II-III lung cancer
  Interventions: Procedure: Open surgery

INTERVENTIONS:
Procedure: VATS — Patients undergo a standard VATS operation for stage II-III lung cancer called a lobectomy.
  Arms: VATS
Procedure: Open surgery — Patients undergo a standard open operation for stage II-III lung cancer called a lobectomy.
  Arms: open surgery

SUMMARY:
For patients with stage I lung cancer, the NCCN guidelines point out that if the patient has no contraindications for anatomy and surgery, as long as it does not violate the standard of tumor treatment and the principle of thoracic surgery, it is highly recommended of VATS or minimally invasive surgery.

Although previous papers seem to have obvious advantages, there is a lack of clinical prospective data from patients with stage II-III lung cancer, and especially in the prevalence of uniportal VATS, there is still no objective analysis of this hypothesis. Therefore, the investigators plan to conduct a randomized, prospective study to compare perioperative complications, postoperative pain, life quality, lung function recovery, tumor-free survival rate, etc., in lobectomy for stage II-III lung cancer patients with VATS and thoracotomy.

DETAILED DESCRIPTION:
Lung cancer is the most common malignant tumor in the world. Surgical treatment is the first and most important treatment for lung cancer. It can completely remove the primary lesions of lung cancer and metastasis of lymph nodes to achieve clinical cure. Opening the chest into the chest allows for an excellent surgical field of view, but it is usually necessary to divide the pectoralis and separate the ribs. To prevent these shortcomings, in the early 1990s, video-assisted thoracoscopic surgery (VATS) was first applied to anatomical pneumonectomy and proved to be safe and feasible. Nowadays, for patients with stage I lung cancer, the NCCN guidelines point out that if the patient has no contraindications for anatomy and surgery, as long as it does not violate the standard of tumor treatment and the principle of thoracic surgery, it is highly recommended of VATS or minimally invasive surgery.

For lung cancer, the benefit of VATS over open surgery is mainly due to the reduction of surgical trauma and the relative maintenance of chest integrity, the reduction of immune function, the reduction of postoperative pain, and the preservation of lung and shoulder function. What's more, the incidence of postoperative complications is reduced, patients recover faster, hospitalization is short, and normal activities are restored early. Although previous papers seem to have obvious advantages, there is a lack of clinical prospective data from patients with stage II-III lung cancer, and especially in the prevalence of uniportal VATS, there is still no objective analysis of this hypothesis.

Therefore, the investigators plan to conduct a randomized, prospective study to compare perioperative complications, postoperative pain, life quality, lung function recovery, tumor-free survival rate, etc., in lobectomy for stage II-III lung cancer patients with VATS and thoracotomy. the investigators would complete the real and effective accumulation of data through strict enrollment, detailed records, and regular follow-up, in order to provide suggestions for the development of new guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of stage II-III non-small cell lung cancer by CT and PET-CT and requiring radical surgery for lung cancer;
2. Age ≥ 18 years.

Exclusion Criteria:

1. palliative surgery;
2. previous thoracic surgery;
3. chest wall resection;
4. Pancoast tumors;
5. reconstruction of carina.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
disease free survival after surgery | 3 years
  Determine if VATS provides a non inferior oncologic control to open Lobectomy, as measure by 3-year progression free survival.

SECONDARY OUTCOMES:
Postoperative pain | 6 month
  Numericrating scale (NRS) is to asses the development of acute and chronic pain after VATS surgery. 11 point numeric rating scale of 0 represented "no pain"and a score of 10 represented "worst pain ".
Quality of life | 6 month
  The EQ5D questionnaire consists of five questions (primary dimensions) about mobility, self-care, usual activities, pain and discomfort, and anxiety and depression, which all have three possible answers ("no problems", "some problems", or "extreme problems"). Additionally, EQ5D includes self-reported overall quality of life as a linear 100 point scale, where 0 is the worst imaginable health state and 100 is the best imaginable health state. EORTC QLQ-C30 is a 30-item questionnaire, from which six functional domains of quality of life (physical function, emotional function, cognitive function, social function, and role function), and nine symptom domains (fatigue, pain, nausea and vomiting, dyspnoea, insomnia, appetite, constipation, diarrhoea, and financial difficulties) can be extracted, as well as an overall score.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided